CLINICAL TRIAL: NCT02843035
Title: A 4-part, Open-label, Multicenter, Multinational Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamic, and Exploratory Efficacy of Venglustat in Combination With Cerezyme in Adult Patients With Gaucher Disease Type 3 With Venglustat Monotherapy Extension
Brief Title: Venglustat in Combination With Cerezyme in Adult Patients With Gaucher Disease Type 3 With Venglustat Monotherapy Extension
Acronym: LEAP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDY13949; U1111-1156-4278 (Registry Identifier: ICTRP); 2023-508646-18 (Registry Identifier: CTIS); 2014-002550-39 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Gaucher Disease Type 1; Gaucher Disease Type 3
MeSH Terms: conditions — Gaucher Disease | interventions — venglustat; imiglucerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (OL) venglustat (Experimental): Administered once a day orally for up to approximately 10 years. Participants will continue their usual dose of Cerezyme during Part 1, Part 2 and Part 3. There is no administration of Cerezyme in Part 4 unless administrated as rescue treatment.
  Interventions: Drug: venglustat (GZ402671); Drug: imiglucerase

INTERVENTIONS:
Drug: venglustat (GZ402671) — Pharmaceutical form: capsule or tablet
  Route of administration: oral
Drug: imiglucerase — Pharmaceutical form: sterile lyophilized product
  Route of administration: intravenous
  Other Names: Cerezyme

SUMMARY:
Part 1: Biomarker evaluation/screening phase

Primary Objectives:

* Evaluate cerebrospinal fluid (CSF) biomarkers in adult Gaucher disease Type 3 (GD3) participants that distinguish GD3 from adult Gaucher disease Type 1 (GD1) participants
* Screen adult GD3 participants who qualify for treatment with venglustat in Parts 2, Part 3, and Part 4 Parts 2 and 3: Combination treatment phases

Primary objectives:

* Evaluate short-term (Part 2) and long-term (Part 3) safety and tolerability of venglustat in combination with Cerezyme in adult GD3 participants
* Evaluate the change in CSF central nervous system (CNS) biomarkers (glucosylceramide [GL-1] and lyso-glucosylceramide [lyso-GL-1]) from adult GD3 participants receiving venglustat in combination with Cerezyme (Part 2 only) Part 4: Extended treatment phase with monotherapy

Primary objectives:

• Evaluate safety and tolerability of venglustat monotherapy in adult GD3 participants who have remained systemically stable on venglustat in combination with Cerezyme Parts 2 and 3: Combination treatment phases

Secondary Objectives:

* Evaluate the pharmacokinetics (PK) of venglustat in adult GD3 participants
* Evaluate the efficacy of venglustat in combination with Cerezyme in systemic disease in adult GD3 participants by assessing spleen volume, liver volume, hemoglobin level and platelet count
* Evaluate the efficacy of venglustat in combination with Cerezyme on neurological function in adult GD3 participants by assessing Ataxia using the Scale for the Assessment and Rating of Ataxia (SARA)
* Evaluate plasma biomarkers (lyso-GL-1 and GL-1) in adult GD3 participants Part 4: Extended treatment phase with monotherapy

Secondary objectives:

* Evaluate the efficacy of venglustat in systemic disease in adult GD3 participants by assessing spleen volume, liver volume, hemoglobin level and platelet count
* Evaluate the efficacy of venglustat on neurological function in adult GD3 participants by assessing Ataxia using the Scale for the Assessment and Rating of Ataxia (SARA)
* Evaluate plasma biomarkers (lyso-GL-1 and GL-1) in adult GD3 participants

DETAILED DESCRIPTION:
The total duration for GD1 participants is 45 days (Part 1), while for GD3 participants the total duration is up to approximately 10 years

ELIGIBILITY:
Inclusion Criteria:

GD3 and GD1 participants must meet the following criteria to be eligible for this study:

* GD1 participant is ≥18 and ≤40 years of age.
* GD3 participant is ≥18 years of age.
* Participant must provide written informed consent prior to any study-related procedures being performed.
* Participant has a clinical diagnosis of Gaucher disease Type 1 (GD1) or Gaucher disease Type 3 (GD3) and documented deficiency of acid beta-glucosidase activity confirming this diagnosis.
* Participant has received ERT (Cerezyme or other ERT; as deemed appropriate by local regulations) for at least 3 years prior to enrollment, on a stable dose for at least 6 months and is within the therapeutic goals defined below, and is deemed clinically stable for at least 1 year by the Investigator.
* Participant has reached Gaucher disease therapeutic goals defined as all of the following to be eligible for this study:

  * Hemoglobin level of ≥11.0 g/dL for females and ≥12.0 g/dL for males.
  * Platelet count ≥100,000/mm3.
  * Spleen volume <10 multiples of normal (MN), or total splenectomy (provided the splenectomy occurred >3 years prior to randomization).
  * Liver volume <1.5 MN.
  * No bone crisis and free of symptomatic bone disease such as bone pain attributable to osteonecrosis and/or pathological fractures within 3 months prior to screening.
* Participant has maintained GD therapeutic goals defined as all of the following to be eligible for entering Part 4 of this study:

  * Hemoglobin level of ≥11.0 g/dL for females and ≥12.0 g/dL for males
  * Platelet count ≥100 000/mm3
  * Spleen volume <10 multiples of normal (MN), or total splenectomy
  * Liver volume <1.5 MN
  * No bone crisis and free of symptomatic bone disease such as bone pain attributable to osteonecrosis and/or pathological fractures within 3 months prior to entering Part 4
* Participant, if female and of childbearing potential, must have a negative pregnancy test [urine beta-human chorionic gonadotropin (β-hCG)] at baseline.
* If participant has a history of seizures, except for myoclonic seizures, they are well controlled under appropriate medication not identified as a strong or moderate inducer or inhibitor of cytochrome P450 (CYP) 3A.
* Participant is willing to abstain from consumption of grapefruit, grapefruit juice, or grapefruit containing products for 72 hours prior to administration of the first dose of venglustat and for the duration of the treatment period.
* Oculomotor apraxia characterized by a horizontal saccade abnormality.
* Female participants of childbearing potential and male participants must be willing to practice true abstinence in line with their preferred and usual lifestyle, or use 2 acceptable effective methods of contraception for the duration of the study and for at least 6 weeks for females and 90 days for males following their last dose of venglustat.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Substrate reduction therapy or chaperone therapy for GD within 6 months prior to enrollment.
* Participant has had a partial or total splenectomy within 3 years prior to randomization.
* Participant is blood transfusion-dependent.
* Prior esophageal varices or liver infarction or current liver enzymes (alanine aminotransferase [ALT]/ aspartate aminotransferase [AST]) or total bilirubin >2 times the upper limit of normal, unless the participant has a diagnosis of Gilbert Syndrome.
* Participant has any clinically significant disease, other than GD, including cardiovascular (congenital cardiac defect, coronary artery disease, valve disease or left sided heart failure; clinically significant arrhythmias or conduction defect), hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic (eg, hypokalemia, hypomagnesemia) or psychiatric disease, other medical conditions, or serious intercurrent illnesses that may preclude participation.
* Participant has renal insufficiency, as defined by an estimated glomerular filtration rate <30 mL/min/1.73m2 at the screening visit.
* Participant has received an investigational product within 30 days prior to enrollment.
* Participant has a history of cancer, with the exception of basal cell carcinoma.
* Participant has myoclonic seizures.
* Participant is pregnant or lactating.
* Participant has, according to World Health Organization (WHO) Grading, a cortical cataract > one-quarter of the lens circumference (Grade cortical cataract-2) or a posterior subcapsular cataract >2 mm (Grade posterior subcapsular cataract-2). Participants with nuclear cataracts will not be excluded.
* Participant requires use of invasive ventilatory support.
* Participant requires use of noninvasive ventilator support while awake for longer than 12 hours daily.
* Participant is unable to receive treatment with Cerezyme due to a known hypersensitivity or is unwilling to receive Cerezyme treatment to ensure maintenance of Gaucher treatment goals.
* Participant is currently receiving potentially cataractogenic medications (corticosteroids, psoralens used in dermatology with ultraviolet light therapy [PUVA], typical antipsychotics, and glaucoma medications) or any medication that may worsen the vision of a participant with cataract (eg, alphaadrenergic glaucoma medications).
* Participant has received strong or moderate inducers or inhibitors of CYP3A within 15 days or 5 half-lives from screening, whichever is longer, prior to enrolment in Part 2. This also includes the consumption of grapefruit, grapefruit juice, or grapefruit containing products within 72 hours of starting venglustat administration in Parts 2 and 3.
* Participant is scheduled for in-patient hospitalization including elective surgery, during the study.
* Participant has had a major organ transplant (e.g., bone marrow or liver).
* Participant, in the opinion of the investigator, is unable to adhere to the requirements of the study or unable to undergo study assessments (e.g., contraindications for magnetic resonance imaging).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | From screening up to end of study, up to approximately 10 years
Assessment of pharmacodynamic (PD) parameter: Lyso-glucosylceramide (lyso-GL1) and glucosylceramide (GL-1) in cerebrospinal fluid (CSF) | From screening through Week 52

SECONDARY OUTCOMES:
Assessment of pharmacodynamic (PD) parameter: Lyso-glucosylceramide (lyso-GL1) and glucosylceramide (GL-1) in plasma | From screening up to end of study, up to approximately 10 years
  Change from baseline in plasma lyso-GL1 and GL1
Assessment of plasma pharmacokinetic parameter: Cmax (Part 2) | Day 1
  Plasma maximum concentration (Cmax)
Assessment of plasma pharmacokinetic parameter: Tmax (Part 2) | Day 1
  Plasma time at Cmax (Tmax)
Assessment of plasma pharmacokinetic parameter: AUC0-24h (Part 2) | Day 1
  Plasma area under the curve (AUC0-24h)
Assessment of plasma pharmacokinetic parameter: Ctrough | Weeks 12 and 39 (Part 2), and on Weeks 78, 104, and 156 (for Part 3)
  Plasma trough concentration (Ctrough)
Assessment of CSF pharmacokinetic parameter: Cmax | Week 4, Week 26, and Week 52
  CSF maximum concentration (Cmax)
Assessment of spleen volume | From screening up to end of study, up to approximately 10 years
  Percent change from baseline in spleen volume assessed by Magnetic Resonance Imaging (MRI)
Assessment of spleen volume (Part 4) | From Week 260 up to end of study, up to approximately 10 years
  Percent change from Part 4 baseline in spleen volume assessed by MRI
Assessment of liver volume | From screening up to end of study, up to approximately 10 years
  Percent change from baseline in liver volume assessed by MRI
Assessment of liver volume (Part 4) | From Week 260 up to end of study, up to approximately 10 years
  Percent change from Part 4 baseline in liver volume assessed by MRI
Assessment of hemoglobin level | From screening up to end of study, up to approximately 10 years
  Change from baseline in hemoglobin level
Assessment of hemoglobin level (Part 4) | From Week 260 up to end of study, up to approximately 10 years
  Change from Part 4 baseline in hemoglobin level
Assessment of platelet level | From screening up to end of study, up to approximately 10 years
  Percent change from baseline in platelet count
Assessment of platelet level (Part 4) | From Week 260 up to end of study, up to approximately 10 years
  Percent change from Part 4 baseline in platelet count
Assessment of Ataxia | From screening up to end of study, up to approximately 10 years
  Ataxia is assessed by using the Scale for the Assessment and Rating of Ataxia (SARA), which consists of 8 items that are related to gait, stance, sitting, speech disturbance, finger-chase test, nose-finger test, fast alternating hand movements and heel-shin slide test. A modified scoring algorithm is used to determine the SARA modified total score from 0 (no ataxia) to 32 (very severe ataxia).
  Change from baseline in SARA modified total score.
Assessment of Ataxia (Part 4) | From Week 260 up to end of study, up to approximately 10 years
  Ataxia is assessed by using the Scale for the Assessment and Rating of Ataxia (SARA), which consists of 8 items that are related to gait, stance, sitting, speech disturbance, finger-chase test, nose-finger test, fast alternating hand movements and heel-shin slide test. A modified scoring algorithm is used to determine the SARA modified total score from 0 (no ataxia) to 32 (very severe ataxia).
  Change from Part 4 baseline in SARA modified total score.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States (3):
  - Yale University School of Medicine Site Number : 840002, New Haven, Connecticut
  - Baylor Institute of Metabolic Diseases Site Number : 840001, Dallas, Texas
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc Site Number : 840003, Fairfax, Virginia
- Investigational Site Number : 276001, Mainz, Germany
- Investigational Site Number : 392001, Minato-ku, Tokyo, Japan
- United Kingdom (2):
  - Investigational Site Number : 826003, Cambridge, Cambridgeshire
  - Investigational Site Number : 826002, Salford, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Schiffmann R, Mengel E, Wallace M, Rochmann C, Turnbull J, Krupnick R, Gwaltney C, Pulikottil-Jacob R, Batsu I, Zheng R, Hamed A. Qualitative Study of the Patient Experience with Venglustat for Gaucher Disease Type 3 in a Phase 2 Open-Label, Multicenter, Multinational Study (LEAP). Adv Ther. 2024 Jul;41(7):2907-2923. doi: 10.1007/s12325-024-02881-2. Epub 2024 May 27. PMID 38802634